CLINICAL TRIAL: NCT02541513
Title: An Open-label Study of Oral Paliparidone for the Treatment of Patients With Co-occurring Opioid and Amphetamine-type Stimulant Dependence
Brief Title: An Open-label Study of Oral Paliparidone for the Treatment of Patients With Co-occurring Opioid and ATS Dependence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Vicknasingam B Kasinather, Dr, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00004494a
Record Dates: First submitted 2015-06-29; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Heroin Dependence; Amphetamine Dependence
Keywords: paliparidone; amphetamine type stimulant dependence
MeSH Terms: conditions — Heroin Dependence; Amphetamine-Related Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paliparidone (Experimental): All patients will begin receiving oral paliperidone 3 mg daily for 3 days followed by an injection of Paliperidone 150 mg injection on Day 8
  Interventions: Drug: paliparidone

INTERVENTIONS:
Drug: paliparidone — All patients will begin receiving oral paliperidone 3 mg daily for three days, beginning on Day 5 of the inpatient phase. All patients will receive an injection of Paliperidone 150 mg injection on Day 8 of the inpatient phase. Patients will receive monthly 150 mg injection for the next 3 months.
  Other Names: invega

SUMMARY:
The proposed study will evaluate the tolerability, acceptability and potential efficacy of paliparidone for the treatment of co-occurring opioid and amphetamine-type stimulant (ATS) dependence. In the proposed clinical trial, all patients will first discontinue illicit opioid and ATS and be inducted onto buprenorphine maintenance treatment (BMT) in the inpatient ward at the department of psychiatry before beginning to receive paliparidone. Tolerability and acceptability will be evaluated by assessing the rates of patient retention during treatment, patient satisfaction with treatment and adverse effects during treatment. The potential efficacy of paliparidone will be evaluated with regard to the primary outcome measure: reductions in illicit ATS use, based on urine toxicology testing and self-report. Secondary outcome measures include treatment retention, reduction in HIV risk behaviors and improvements in functional status.

DETAILED DESCRIPTION:
Malaysia has been struggling in fighting drug addiction in the country (NADI, 2005). Opioids predominantly heroin and morphine and ATS (Chawarski et al, 2006). dependence are the primary drugs of abuse for most drug users in Malaysia There are more than 300,000 registered drug users in Malaysia, most are opioid dependent and current intravenous drug users (IVDU). Drug abuse comes together with other medical and social problems, as 25-30% of IVDU are infected with HIV; and IVDU accounts for 70% of HIV infections in Malaysia. There are more than 90, 000 registered HIV positives between 1986 and 2010. (National Anti-Drug Agency of Malaysia, 2010).

Over the past decade, amphetamine-type stimulant (ATS) has also emerged as a major drug problem. Globally, ATS is now the second most commonly used illicit drug type and is more widely used than heroin. ATS abuse is especially prevalent and problematic in the Asian region, where ATS production, use, drug seizures, and demand for treatment have continued to increase. Injection of methamphetamine has been reported in Malaysia (Chawarski et al, 2006) and other south-east Asian countries (McKetin, 2008). In the most recent survey of out-of-treatment heroin IVDU in cities across Malaysia, more than 60% report current ATS use, and 29% inject ATS (Chawarski et al, 2012).

ATS use is associated with increased HIV transmission behavioral risks. The connection of heroin, methamphetamine and HIV in Malaysia is well documented (Chawarski et al, 2006). Increased needle sharing and risky sexual behaviors lead to increased prevalence of HIV infection. ATS use exacerbates HIV transmission risk through a number of mechanisms: ATS users report engaging in more frequent and more risky sexual behaviors while using ATS and in more frequent needle sharing. ATS is also associated with impairments of mood and executive functioning that may persist for prolonged periods and may contribute to relapse to drug use, thus all other problems.

Drug abuse has been a major problem in Kelantan for the past several decades (Suarn & NorAdam,1993) and ATS has been gaining momentum over the past decade. The number of individuals arrested annually for ATS in Kelantan increased over the past 5 years from 2900 in 2007 to 5300 in 2010. For the past 5 years, Kelantan has also led Malaysia in having the highest population prevalence of HIV infection, at 47 per 100,000 in 2008, nearly 4 times the prevalence reported for the rest of Malaysia. Kelantan also has the highest number of women with HIV in Malaysia with more than 1200 reported in 2008, suggesting that HIV is making the transition to the general population. A large proportion of treatment seeking drug users in Kelantan are HIV positives and are susceptible to high mortality (JKNK, 2012).

Paliperidone, the primary active metabolite of risperidone, is a long-acting atypical neuroleptic (antipsychotic) medication. It blocks dopamine 2 (D2) receptors and serotonin 2A receptors and acts as an alpha2 antagonist. Blockade of the D2 receptors may reduce the reinforcing effects of ATS or other stimulants; blockade of the serotonin 2A receptor leads to increased DA release in the prefrontal cortex and motor regions and may thus improve cognitive performance and mood and reduce motor impairments associated with blockade of D2 receptors; and alpha2 antagonist actions may provide antidepressant effects.

Paliperidone's potential efficacy for treating ATS dependence was suggested both by its potential for blocking or attenuating the rewarding effects of ATS use and by its potential for improving cognitive functioning in patients recovering from ATS dependence. An open label pilot study of oral risperidone for the treatment of methamphetamine dependence provided preliminary evidence for the safety, tolerability and potential efficacy of risperidone. Risperidone was generally well-tolerated and associated with decreased methamphetamine use and improvements in fine motor function and mood. A subsequent open trial of injectable ripseridone found that injectable risperidone was associated with reductions in methamphetamine use and improvements in verbal memory.

However to date there have been no published replication studies or studies of paliperidone for treating ATS dependence in other populations and setting. This proposed pilot study of paliperidone for the treatment of ATS dependence would extend this work and provide specific data regarding the tolerability and efficacy of paliperidone in opioid-agonist maintained patients with co-occurring ATS and opioid dependence (COATS).

In addition to detoxification and treatment medications, a manual-guided educational drug and HIV risk reduction counseling (EDRC) will be provided to all participants. EDRC provides education about medical understanding of opioid and ATS addiction, highly effective strategies used in successful drug recovery efforts, medical and other harmful consequences of drug use including HIV and other infectious disease transmission, as well as about effective prevention of all negative consequences of illicit drug use (Chawarski et al, 2008). It helps patient to remain in treatment, adhere to prescribed medications, abstain from or reduce illicit opioid and ATS use and HIV risk behaviors, and make life-style changes fostering sustained recovery. It also teaches basic cognitive and behavioral coping skills that increase the patients' chances to reach sustained and prolonged recovery from drugs. For HIV positive patients, EDRC encourages patients to attend the HIV clinic and adhere to monitoring, medication, and other treatment recommendations. EDRC will be provided by trained and supervised nursing personnel, drug counselors, or therapists. It will be offered in individual format with the frequency ranging from 3 times per week during detoxification to once per week during the outpatient phase of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV criteria for both opioid and ATS dependence, as assessed by the Structured Clinical Interview for DSM (SCID)
2. Active COATS dependence as documented by ATS and opioid-positive urine tests and a report of at least 2 or more days per week of ATS use over the past month.
3. Age 18 - 65 years old

Exclusion Criteria:

1. Liver enzymes greater than 3 times the upper limit of normal or evidence of liver failure or acute hepatitis.
2. Having serious medical or psychiatric illnesses: (including current psychotic disorder, major depression, suicidal or homicidal ideations) or taking medications to treat depression or psychosis.
3. Refused informed consent or inability to understand the protocol or assessment questions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in illicit ATS use | 18 weeks
  This will be measured from baseline over time during treatment, based on urine toxicology testing and self-report

SECONDARY OUTCOMES:
Reductions in sexual and drug-related HIV risk behaviors | 18 weeks
  Measured by monthly self-report assessments using a questionnaire
Measure improvements in neuropsychological functioning, | 18 weeks
  Measured by repeated assessments of neuropsychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Vicknasingam Kasinather, PhD, Principal Investigator — University Science Malaysia
Locations (1):
- University Science Malaysia, Kota Bharu, Kelantan, Malaysia